CLINICAL TRIAL: NCT04585204
Title: Comparison of the Detection Rates of 50 Gr-100 Gr OGTT and 75 Gr OGTT That Require Medical Treatment of GDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E1-20-800
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Gestational Diabetes; Glucose Intolerance During Pregnancy
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50 gr-100 gr OGTT (Active Comparator): patients are tested firstly by 50 gr OGTT after that if necessary by 100 gr OGTT
  Interventions: Diagnostic Test: Oral glucose tolerance test
- 75 gr OGTT (Active Comparator): patients are tested by 75 gr OGTT
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — Oral glucose tolerance test

SUMMARY:
Both 50 gr OGTT-100 gr OGTT and 75 gr OGTT are used for detecting gestational diabetes mellitus. Two approaches are approved by obstetricians. With this study, we aim to compare the gestational diabetes mellitus detection rate of these different tests.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

Exclusion Criteria:

* Already diagnosed by diabetes mellitus
* Multiple pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2282 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
the difference of GDM detection rate of 50 gr- 100 gr OGTT and 75 gr OGTT | one year
  to determine the ideal diagnostic test

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided